CLINICAL TRIAL: NCT06655935
Title: Novel Modified Technique for Transcatheter Closure of Secundum Atrial Septal Defect: A Single Center Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Nouran Mostafa Mansour, dr, Egyptian Biomedical Research Network
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 36264PR84/2/23
Record Dates: First submitted 2024-10-16; First posted 2024-10-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Atrial Septal Defect (ASD)
Keywords: atrial septal defects; transcatheter closure; modified technique
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 44 patients with ASD who underwent the ordinary transcatheter closure technique using ASO. (Active Comparator): The dilator of the Amplatzer delivery sheath of the Amplatzer™ Septal Occluders ASO is advanced over stiff wire into the pulmonary veins
  Interventions: Procedure: Ordinary Transcatheter ASD closure
- 36 patients with ASD who underwent the modified transcatheter closure technique using ASO (Experimental): Amplatzer delivery sheath of the Amplatzer™ Septal Occluders ASO is advanced over the multipurpose catheter to the left atrial cavity
  Interventions: Procedure: modified transcatheter ASD closure

INTERVENTIONS:
Procedure: Ordinary Transcatheter ASD closure — deploying the Amplatzer delivery system of the Amplatzer™ Septal Occluders ASO inside the left atrial cavity over stiff wire into the pulmonary veins
  Arms: 44 patients with ASD who underwent the ordinary transcatheter closure technique using ASO.
Procedure: modified transcatheter ASD closure — deploying the Amplatzer delivery system of the Amplatzer™ Septal Occluders ASO over the multipurpose catheter inside the left atrial cavity which might help in the shortage of the duration & the cost of the procedure with less complication rate
  Arms: 36 patients with ASD who underwent the modified transcatheter closure technique using ASO

SUMMARY:
Transcatheter closure of secundum atrial septal defects is widely approved worldwide, yet it still has multiple risks like perforation and radiation exposure. In this study, we proposed a modified rapid method for closure of secundum atrial septal defects, to avoid material manipulation inside your heart and decrease complication rate.

DETAILED DESCRIPTION:
Delivery sheath can be advanced over multipurpose catheter instead of stiff wire

ELIGIBILITY:
Inclusion Criteria:

* Any patient with ostium secundum ASD & RV volume overload

Exclusion Criteria:

* Any other type of atrial septal defects Any other associated congenital anomaly

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
recording any complication during transcatheter secundum atrial septal defect closure | during the procedure
  stiff wire can cause perforation or arrhythmias

SECONDARY OUTCOMES:
assess the duration of the procedure and if this affects the cost of the procedure by any means | during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Raghda El sheikh, professor, Study Director — Cardiology departement-Tanta University hospital
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
because of the confidentiality of the patients data